CLINICAL TRIAL: NCT06181695
Title: Intranasal Sufentanil for Analgesia of Severe Sickle Cell Vaso-occlusive Pain Crisis in the Pediatric Emergency Department: a Double Blind Randomized Versus Placebo Controlled Trial
Brief Title: Intranasal Sufentanil for Analgesia of Severe Sickle Cell Vaso-occlusive Pain Crisis in the Pediatric
Acronym: INVOPE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP211035
Record Dates: First submitted 2023-11-15; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Vaso-occlusive Crisis
MeSH Terms: conditions — Vaso-Occlusive Crises | interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sufentanil IN + Morphine IV (Experimental): Intranasal Sufentanil + IV morphine:
  Interventions: Drug: Sufentanil
- Placebo IN + Morphine IV (Placebo Comparator): Placebo of Sufentanil administered intranasally (IN) . One single administration +IV morphine similar to the experimental arm:
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Sufentanil — Administration of intranasal sufentanil
  Other Names: sufentanil IN + morphine IV

SUMMARY:
Sickle cell disease (SCD) is characterized by an abnormal hemoglobin, the main protein in the red blood cell. From the first months of life, acute obstruction of the vessels of the microcirculation manifests as intense and unpredictable recurrent episodes of severe pain. In the Emergency Department (ED), patients presenting with a vaso-occlusive crisis (VOC) required a rapid evaluation and administration of pain relief therapies and hydration.

this strategy is based on an intranasal (IN) administration of Sufentanil at the initial management of children with VOC, followed by morphine intravenous (IV) relay as soon as possible, compared to the usual care procedure with IV morphine as soon as possible.

The hypothesis is that the use of this IN opioid at the beginning of the management of children with VOC can reduce the time before being pain relieved. Indeed, the IN administration make it easier and faster to administer.

DETAILED DESCRIPTION:
Sufentanil is a powerful opioid analgesic used intravenously by emergency physicians for the sedation of intensive care, intubated and ventilated patients. It is therefore already present in the pharmacopoeia of emergencies. As the duration of action of inztranasal Sufentanil is too short to completely replace the IV morphine, a very promising approach would be to use it during the initial phase of the management of severe pain in children with painful sickle cell crisis while waiting for a venous access.

The INVOPE trial is a phase III trial evaluating the intranasal sufentanil in sickle cell disease children with severe VOC.

The INVOPE trial is a randomized controlled, multicenter, double blind, two parallel-group in a 1:1 ratio, placebo-controlled superiority trial comparing the analgesic efficacy of the sufentanil IN + standard care IV morphine / versus placebo IN + IV morphine as soon as possible.

Children will be randomized in two groups:

* Experimental group: IN Sufentanil procedure with IV administration of morphine as soon as possible
* Control group : IN placebo IN procedure with IV administration of morphine as soon as possible

The objective of this trial is to compare a procedure consisting in IN Sufentanil followed by IV morphine, when compared to IN placebo followed by IV morphine alone, in children with severe vaso-occlusive crisis.

ELIGIBILITY:
Inclusion Criteria:

At inclusion visit:

* Sickle-cell disease = Hemoglobin SS or SC or Sß-thalassemia
* Age < 18 years old
* Weight > 10 kgs
* Registered with the social security scheme (or State Medical Aid - AME) or his/her beneficiaries
* Informed consent of the holder (s) of the exercise of parental authority
* Age < 18 years old

At randomisation visit

* Presenting to the ED with vaso-occlusive crisis: migratory bone pain, which may occur in the limbs, spine, thorax, pelvis, skull; or crisis known as such by the patient.
* Severe pain determined at triage, defined as:

  * EVENDOL ≥ 10/15 in children aged 0-8 years or
  * NRS-11 ≥ 7/10 in children aged 8 years to less than 18 years
* Informed consent of the holder (s) of the exercise of parental authority signed at inclusion visit

Exclusion Criteria:

* At inclusion visit

  * Known cirrhosis
  * End-stage renal disease requiring kidney dialysis
  * Known hypersensitivity or contraindication to sufentanil or any of the excipients
  * Contraindication to morphine
  * Facial malformation, epistaxis, blocked or traumatised nose
  * Severe asthma
  * Patient's or parent's refusal to participate
  * Participation in another interventional trial
  * Parents who do not speak French

At randomization visit

* Known cirrhosis
* End-stage renal disease requiring kidney dialysis
* Known hypersensitivity or contraindication to sufentanil or any of the excipients
* Contraindication to morphine
* Facial malformation, epistaxis, blocked or traumatised nose
* Severe asthma
* Patient's or Parent's refusal to participate or withdrawal of parental consent
* Participation in another interventional trial
* Patient has already been randomised to the INVOPE trial during a previous VOC
* Strong opioids received <6 hours (morphine, oxycodone, hydromorphone, fentanyl, sufentanil, nalbuphine)
* Respiratory failure (tachypnea; bradypnea; paradoxical breathing; grunting; head-bobbing; nasal flaring; retractions (subcostal, suprasternal, intercostal, sternal))
* Oxygen saturations below 95% on initial assessment
* Pneumonia requiring oxygen therapy
* Hemodynamic disorders: tachycardia, hypotension
* Altered conscious state as defined by a Glasgow Coma score less than 15
* Positive urinary pregnancy test for woman of childbearing potential (postpubertal female with sexual activity)
* Nasal or sinus surgery within 6 months before randomisation
* High fever > 39°C
* Sign of intolerance of acute anaemia
* Description by the patient (or the parents) of the unusual nature of the attack

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 182 (Estimated)
Dates: Start 2024-05-02 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-05-29 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the Efficacy of Intra-nasal Sufentanil for Analgesia of Vaso-occlusive Crisis in Sickle-cell in children | at 30 minutes
  efficacy of the analgesia at 30 minutes after IN injection, in children with SCD presenting to the pediatric ED with a severe VOC with Pain relief is defined as EVENDOL score ≤ 5/15 or NRS-11 score ≤ 3/10

SECONDARY OUTCOMES:
Proportion of children relieved (EVENDOL ≤ 5/15 or NRS-11 ≤ 3/10) at 10, 20, 40, 50 and 60 minutes after the IN injection inclusion | at 60 minutes
  Proportion of children relieved (EVENDOL ≤ 5/15 or NRS-11 ≤ 3/10) at 10, 20, 40, 50 and 60 minutes after the IN injection inclusion
Proportion of children with a moderate pain (EVENDOL ≤ 9/15 or NRS-11 ≤ 6/10) at 10, 20, 30, 40, 50 and 60 minutes after the IN injection | EVENDOL ≤ 5/15 or NRS-11 ≤ 3/10 at 10, 20, 40, 50 and 60 minutes
  Proportion of children relieved (EVENDOL ≤ 5/15 or NRS-11 ≤ 3/10) at 10, 20, 40, 50 and 60 minutes after the IN spray;
To demonstrate that {IN Sufentanil +IV morphine(as a standard of care)} procedure, when compared to {IN Placebo + IV morphine (as a standard of care)} procedure, is able to decrease the level of morphine consumption | from randomisation to 60 minutes after
  Morphine consumption (mg). Assessed morphine consumption after treatment initiation, until 60 minutes
To demonstrate the safety of the {IN Sufentanil +IV morphine} procedure, when compared to {IN Placebo + IV morphine } procedure, that is an absence of increase rate of hemodynamic and non-hemodynamic side effects of opiace | until 4 hours after the IN injection
  Rates of hypotension, hypoxia, bradycardia, respiratory distress, headache, nausea, vomiting, sleepiness and itchiness until 4 hours after the IN injection
To evaluate the safety of all children aged 0-18 years | From randomisaton to 4 hours after
  This outcome is defined by the proportion of patients with at least one adverse events during the medical care, until 4 hours after treatment initiatio
To demonstrate that the {IN Sufentanil +IV morphine (as a standard of care)} procedure, when compared to {IN Placebo + IV morphine (as a standard of care)} procedure, is able to improve the management of a VOC episode | after 4 hours of randomisation
  Rate of admission after the ED visit
To demonstrate that the {IN Sufentanil +IV morphine (as a standard of care)} procedure, when compared to {IN Placebo + IV morphine(as a standard of care)} procedure, is able to decrease the proportion of VOC complications | at hospital discharg, after 4 hours after randomisation
  Rate of Acute chest syndrome: at hospital discharge Rate of admission in ICU, invasive ventilation, non-invasive ventilation, oxygene therapy: at hospital discharge Rate of Transfusion: at hospital discharge Rate of death: at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Camille AUPIAIS, Pre, Principal Investigator — Assistance Publique des Hopitaux de Paris

REFERENCES:
- [Background] Prise en charge de la drépanocytose chez l'enfant et l'adolescent. Haute Autorité de Santé. Accessed March 3, 2021. https://www.has-sante.fr/jcms/c_272479/fr/prise-en-charge-de-la-drepanocytose-chez-l-enfant-et-l-adolescent
- [Background] Yawn BP, Buchanan GR, Afenyi-Annan AN, Ballas SK, Hassell KL, James AH, Jordan L, Lanzkron SM, Lottenberg R, Savage WJ, Tanabe PJ, Ware RE, Murad MH, Goldsmith JC, Ortiz E, Fulwood R, Horton A, John-Sowah J. Management of sickle cell disease: summary of the 2014 evidence-based report by expert panel members. JAMA. 2014 Sep 10;312(10):1033-48. doi: 10.1001/jama.2014.10517. PMID 25203083
- [Background] Gonzalez ER, Bahal N, Hansen LA, Ware D, Bull DS, Ornato JP, Lehman ME. Intermittent injection vs patient-controlled analgesia for sickle cell crisis pain. Comparison in patients in the emergency department. Arch Intern Med. 1991 Jul;151(7):1373-8. PMID 2064488
- [Background] Dampier CD, Smith WR, Wager CG, Kim HY, Bell MC, Miller ST, Weiner DL, Minniti CP, Krishnamurti L, Ataga KI, Eckman JR, Hsu LL, McClish D, McKinlay SM, Molokie R, Osunkwo I, Smith-Whitley K, Telen MJ; Sickle Cell Disease Clinical Research Network (SCDCRN). IMPROVE trial: a randomized controlled trial of patient-controlled analgesia for sickle cell painful episodes: rationale, design challenges, initial experience, and recommendations for future studies. Clin Trials. 2013 Apr;10(2):319-31. doi: 10.1177/1740774513475850. PMID 23539110
- [Background] Treadwell MJ, Bell M, Leibovich SA, Barreda F, Marsh A, Gildengorin G, Morris CR. A Quality Improvement Initiative to Improve Emergency Department Care for Pediatric Patients with Sickle Cell Disease. J Clin Outcomes Manag. 2014 Feb;21(2):62-70. PMID 26412961
- [Background] Shenoi R, Ma L, Syblik D, Yusuf S. Emergency department crowding and analgesic delay in pediatric sickle cell pain crises. Pediatr Emerg Care. 2011 Oct;27(10):911-7. doi: 10.1097/PEC.0b013e3182302871. PMID 21960091
- [Background] Kavanagh PL, Sprinz PG, Wolfgang TL, Killius K, Champigny M, Sobota A, Dorfman D, Barry K, Miner R, Moses JM. Improving the Management of Vaso-Occlusive Episodes in the Pediatric Emergency Department. Pediatrics. 2015 Oct;136(4):e1016-25. doi: 10.1542/peds.2014-3470. Epub 2015 Sep 21. PMID 26391933
- [Background] Brandow AM, Nimmer M, Simmons T, Charles Casper T, Cook LJ, Chumpitazi CE, Paul Scott J, Panepinto JA, Brousseau DC. Impact of emergency department care on outcomes of acute pain events in children with sickle cell disease. Am J Hematol. 2016 Dec;91(12):1175-1180. doi: 10.1002/ajh.24534. Epub 2016 Sep 3. PMID 27517842
- [Background] Mathias MD, McCavit TL. Timing of opioid administration as a quality indicator for pain crises in sickle cell disease. Pediatrics. 2015 Mar;135(3):475-82. doi: 10.1542/peds.2014-2874. Epub 2015 Feb 9. PMID 25667245
- [Background] Galeotti C, Courtois E, Carbajal R. How French paediatric emergency departments manage painful vaso-occlusive episodes in sickle cell disease patients. Acta Paediatr. 2014 Dec;103(12):e548-54. doi: 10.1111/apa.12773. Epub 2014 Oct 2. PMID 25130719
- [Background] Corrigan M, Wilson SS, Hampton J. Safety and efficacy of intranasally administered medications in the emergency department and prehospital settings. Am J Health Syst Pharm. 2015 Sep 15;72(18):1544-54. doi: 10.2146/ajhp140630. PMID 26346210
- [Background] Dale O. Intranasal administration of opioids/fentanyl - Physiological and pharmacological aspects. European Journal of Pain Supplements. 2010;4(3):187-190. doi:10.1016/j.eujps.2010.06.001
- [Background] Dale O, Hjortkjaer R, Kharasch ED. Nasal administration of opioids for pain management in adults. Acta Anaesthesiol Scand. 2002 Aug;46(7):759-70. doi: 10.1034/j.1399-6576.2002.460702.x. PMID 12139528
- [Background] Wolfe TR, Braude DA. Intranasal medication delivery for children: a brief review and update. Pediatrics. 2010 Sep;126(3):532-7. doi: 10.1542/peds.2010-0616. Epub 2010 Aug 9. PMID 20696726
- [Background] Helmers JH, Noorduin H, Van Peer A, Van Leeuwen L, Zuurmond WW. Comparison of intravenous and intranasal sufentanil absorption and sedation. Can J Anaesth. 1989 Sep;36(5):494-7. doi: 10.1007/BF03005373. PMID 2529048
- [Background] Haynes G, Brahen NH, Hill HF. Plasma sufentanil concentration after intranasal administration to paediatric outpatients. Can J Anaesth. 1993 Mar;40(3):286. doi: 10.1007/BF03037044. No abstract available. PMID 8467552
- [Background] Nielsen BN, Friis SM, Romsing J, Schmiegelow K, Anderson BJ, Ferreiros N, Labocha S, Henneberg SW. Intranasal sufentanil/ketamine analgesia in children. Paediatr Anaesth. 2014 Feb;24(2):170-80. doi: 10.1111/pan.12268. Epub 2013 Oct 1. PMID 24118506
- [Background] Murphy A, O'Sullivan R, Wakai A, Grant TS, Barrett MJ, Cronin J, McCoy SC, Hom J, Kandamany N. Intranasal fentanyl for the management of acute pain in children. Cochrane Database Syst Rev. 2014 Oct 10;2014(10):CD009942. doi: 10.1002/14651858.CD009942.pub2. PMID 25300594
- [Background] Lemoel F, Contenti J, Cibiera C, Rapp J, Occelli C, Levraut J. Intranasal sufentanil given in the emergency department triage zone for severe acute traumatic pain: a randomized double-blind controlled trial. Intern Emerg Med. 2019 Jun;14(4):571-579. doi: 10.1007/s11739-018-02014-y. Epub 2019 Jan 1. PMID 30600526
- [Background] Setlur A, Friedland H. Treatment of pain with intranasal fentanyl in pediatric patients in an acute care setting: a systematic review. Pain Manag. 2018 Sep 1;8(5):341-352. doi: 10.2217/pmt-2018-0016. Epub 2018 Oct 3. PMID 30278812
- [Background] Hronova K, Pokorna P, Posch L, Slanar O. Sufentanil and midazolam dosing and pharmacogenetic factors in pediatric analgosedation and withdrawal syndrome. Physiol Res. 2016 Dec 21;65(Suppl 4):S463-S472. doi: 10.33549/physiolres.933519. PMID 28006928
- [Background] Bayrak F, Gunday I, Memis D, Turan A. A comparison of oral midazolam, oral tramadol, and intranasal sufentanil premedication in pediatric patients. J Opioid Manag. 2007 Mar-Apr;3(2):74-8. doi: 10.5055/jom.2007.0043. PMID 17520986
- [Background] Crellin D, Ling RX, Babl FE. Does the standard intravenous solution of fentanyl (50 microg/mL) administered intranasally have analgesic efficacy? Emerg Med Australas. 2010 Feb;22(1):62-7. doi: 10.1111/j.1742-6723.2010.01257.x. PMID 20152004
- [Background] Borland M, Jacobs I, King B, O'Brien D. A randomized controlled trial comparing intranasal fentanyl to intravenous morphine for managing acute pain in children in the emergency department. Ann Emerg Med. 2007 Mar;49(3):335-40. doi: 10.1016/j.annemergmed.2006.06.016. Epub 2006 Oct 25. PMID 17067720
- [Background] Sin B, Jeffrey I, Halpern Z, Adebayo A, Wing T, Lee AS, Ruiz J, Persaud K, Davenport L, de Souza S, Williams M. Intranasal Sufentanil Versus Intravenous Morphine for Acute Pain in the Emergency Department: A Randomized Pilot Trial. J Emerg Med. 2019 Mar;56(3):301-307. doi: 10.1016/j.jemermed.2018.12.002. Epub 2019 Jan 9. PMID 30638644
- [Background] Fantacci C, Fabrizio GC, Ferrara P, Franceschi F, Chiaretti A. Intranasal drug administration for procedural sedation in children admitted to pediatric Emergency Room. Eur Rev Med Pharmacol Sci. 2018 Jan;22(1):217-222. doi: 10.26355/eurrev_201801_14120. PMID 29364490
- [Background] Chiaretti A, Barone G, Rigante D, Ruggiero A, Pierri F, Barbi E, Barone G, Riccardi R. Intranasal lidocaine and midazolam for procedural sedation in children. Arch Dis Child. 2011 Feb;96(2):160-3. doi: 10.1136/adc.2010.188433. Epub 2010 Oct 27. PMID 21030365
- [Background] Inthavong K, Fung MC, Yang W, Tu J. Measurements of droplet size distribution and analysis of nasal spray atomization from different actuation pressure. J Aerosol Med Pulm Drug Deliv. 2015 Feb;28(1):59-67. doi: 10.1089/jamp.2013.1093. Epub 2014 Jun 10. PMID 24914675
- [Background] Barrett MJ, Cronin J, Murphy A, McCoy S, Hayden J, an Fhaili S, Grant T, Wakai A, McMahon C, Walsh S, O'Sullivan R. Intranasal fentanyl versus intravenous morphine in the emergency department treatment of severe painful sickle cell crises in children: study protocol for a randomised controlled trial. Trials. 2012 May 30;13:74. doi: 10.1186/1745-6215-13-74. PMID 22647439